CLINICAL TRIAL: NCT04902950
Title: Role of Tranexamic Acid (TXA) in the Reduction of Post-operative Hematoma and Seroma in Patients Undergoing Panniculectomy or Abdominoplasty, a Pilot Study.
Brief Title: TXA in the Reduction of Post-Op Hematoma and Seroma in Patients Undergoing Panniculectomy or Abdominoplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Logistics
Sponsor: The Reading Hospital and Medical Center (Other)
Responsible Party: Principal Investigator, Amir Behnam, MD FACS Chief, Division of Plastic Surgery, The Reading Hospital and Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB 003-20
Record Dates: First submitted 2021-05-10; First posted 2021-05-26 (Actual); Results first posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Panniculectomy; Abdominoplasty
Keywords: Panniculectomy; Abdominoplasty; Tranexamic acid
MeSH Terms: interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study will be double-blinded. Participating patients will be randomized to receive normal saline (control group) or tranexamic acid (study population) on the day of surgery by the pharmacist. Normal saline is the current standard of care.
  Each group will have 10 participants. Group 1 will undergo application of three normal saline soaked lap sponges to the surgical site. Group 2 will undergo application of three TXA soaked lap sponges to the surgical site. The lap sponges will be removed after three minutes and measurements will be taken for the study.
  After discharge, post-operative drain output will be monitored and recorded by the patient on a provided drain documentation sheet. This does not differ from the current standard of care regarding drain output recordings.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization of the patient is performed by the Pharmacist and entered into REDCap. Access to Patient Group and distributed drug (saline vs TXA) is restricted to the Pharmacist and the Study Coordinator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Placebo Comparator): The solution of saline will be placed into a sterile bowl in the operating area and three lap sponges will be placed in the solution at the beginning of the procedure. Group 1 will undergo application of three normal saline soaked lap sponges to the surgical site. The lap sponges will be removed after three minutes and measurements will be taken for the study.
  Interventions: Drug: Saline
- Group 2 (Experimental): The solution of Tranexamic Acid (TXA) will be placed into a sterile bowl in the operating area and three lap sponges will be placed in the solution at the beginning of the procedure. Group 2 will undergo application of three (TXA) soaked lap sponges to the surgical site. The lap sponges will be removed after three minutes and measurements will be taken for the study.
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — After the abdominal skin and subcutaneous tissue is raised, the area will be irrigated, and hemostasis achieved using electrocautery. These steps are currently preformed with every panniculectomy. The Tranexamic acid soaked lap sponges will be unfolded and placed beneath the two lateral portions as well as the central area of the flap for 3 minutes. The lap sponges will not be "rung out" prior to placement. The surface area under the flap will be measured from the xiphoid process to the pubis, from the Xiphoid process to each anterior superior iliac spine (ASIS) and across from one ASIS to the other. These measurements will be used to calculate the surface area under the flap. These measurements will only be used in data collection and do not affect the principle aim of the study. The remainder of the surgical procedure will be the same for each patient.
  Other Names: TXA
  Arms: Group 2
Drug: Saline — After the abdominal skin and subcutaneous tissue is raised, the area will be irrigated, and hemostasis achieved using electrocautery. These steps are currently preformed with every panniculectomy. The saline soaked lap sponges will be unfolded and placed beneath the two lateral portions as well as the central area of the flap for 3 minutes. The lap sponges will not be "rung out" prior to placement. The surface area under the flap will be measured from the xiphoid process to the pubis, from the Xiphoid process to each anterior superior iliac spine (ASIS) and across from one ASIS to the other. These measurements will be used to calculate the surface area under the flap. These measurements will only be used in data collection and do not affect the principle aim of the study. The remainder of the surgical procedure will be the same for each patient.
  Arms: Group 1

SUMMARY:
The purpose of this study is to study the use of a drug, tranexamic acid (TXA) to decrease bleeding and fluid collections in patients undergoing excision of excess lower abdominal skin and soft tissue, otherwise known as a panniculectomy. The use of TXA in this study is experimental. TXA is a medication currently used in many surgical subspecialties to control bleeding. TXA is approved by the FDA as a medication taken by mouth for the treatment of heavy menstrual bleeding and as an injection in patients with hemophilia for short-term use (two to eight days) to reduce or prevent hemorrhage and reduce the need for replacement therapy during and following tooth extraction.

The use of TXA in this study is experimental, which means it is not approved by the FDA for topical use in decreasing bleeding during and after surgery. The results of this study will help the researchers determine if TXA is effective in decreasing blood loss following surgery. If effective, researchers hope this will result in earlier removal of post-operative drains leading to faster return to work or social activities

DETAILED DESCRIPTION:
Participants consented to take part in this study will be assigned by chance to receive either placebo (Group 1) or TXA (Group 2) during the surgical procedure. This study will be double-blinded, in that neither the patient nor the surgeon will know to which treatment, (placebo vs. TXA) that the patient will receive. Participating patients will be randomized to receive normal saline (control group) or tranexamic acid (study population) on the day of surgery by the pharmacist. Normal saline is the current standard of care. Double blinding ensures that the researcher or the patient's opinion does not influence study results, however this information is available from the pharmacy in the event of any complications.

Each group will have 10 participants. The solution of either saline or TXA will be placed into a sterile bowl in the operating area and three lap sponges will be placed in the solution at the beginning of the procedure. Group 1 will undergo application of three normal saline soaked lap sponges to the surgical site. Group 2 will undergo application of three TXA soaked lap sponges to the surgical site. The lap sponges will be removed after three minutes and measurements will be taken for the study.

After discharge, post-operative drain output will be monitored and recorded by the patient on a provided drain documentation sheet. This does not differ from the current standard of care regarding drain output recordings. All patients who receive a post-surgical drain are asked to document output. All patients will be educated on routine drain care and recording drain output.

Patients will not need to undergo any extra medical tests, medical procedures or doctor visits if they decide to join the study. Patient participation in the study begins upon signature of the consent form and is expected to last no more than 8 weeks following the patient's surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

• Patients undergoing panniculectomy or abdominoplasty.

Exclusion Criteria:

* Prisoners
* Pregnant or nursing women
* Persons under the age of 18
* Preexisting coagulopathy
* Preexisting ongoing venous or arterial thrombosis
* History of cerebral vascular accident
* History of uncontrolled seizure disorder
* Documented administration of daily antiplatelet or anticoagulation (e.g. acetylsalicylic acid ,Non-steroidal anti-inflammatory drugs , Warfarin)
* Documented allergic reaction to tranexamic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Behnam, MD, Principal Investigator — Reading Hospital
Locations (1):
- Reading Hospital, West Reading, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ker K, Beecher D, Roberts I. Topical application of tranexamic acid for the reduction of bleeding. Cochrane Database Syst Rev. 2013 Jul 23;2013(7):CD010562. doi: 10.1002/14651858.CD010562.pub2. PMID 23881695
- [Background] Maj Richard Reed, RAMC, LtCol Tom Woolley, RAMC Continuing Education in Anaesthesia Critical Care & Pain, Volume 15, Issue 1, February 2015, Pages 32-37, https://doi.org/10.1093/bjaceaccp/mku009 Published: 30 May 2014
- [Background] Masoomi H, Rimler J, Wirth GA, Lee C, Paydar KZ, Evans GRD. Frequency and risk factors of blood transfusion in abdominoplasty in post-bariatric surgery patients: data from the nationwide inpatient sample. Plast Reconstr Surg. 2015 May;135(5):861e-868e. doi: 10.1097/PRS.0000000000001161. PMID 25919268
- [Background] Jimenez JJ, Iribarren JL, Lorente L, Rodriguez JM, Hernandez D, Nassar I, Perez R, Brouard M, Milena A, Martinez R, Mora ML. Tranexamic acid attenuates inflammatory response in cardiopulmonary bypass surgery through blockade of fibrinolysis: a case control study followed by a randomized double-blind controlled trial. Crit Care. 2007;11(6):R117. doi: 10.1186/cc6173. PMID 17988379
- [Background] Ausen K, Fossmark R, Spigset O, Pleym H. Randomized clinical trial of topical tranexamic acid after reduction mammoplasty. Br J Surg. 2015 Oct;102(11):1348-53. doi: 10.1002/bjs.9878. PMID 26349843
- [Background] Rohrich RJ, Cho MJ. The Role of Tranexamic Acid in Plastic Surgery: Review and Technical Considerations. Plast Reconstr Surg. 2018 Feb;141(2):507-515. doi: 10.1097/PRS.0000000000003926. PMID 28938364

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Full Range); unit: years] | 39 [36 to 46] | 46 [37 to 58] | 43 [36 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9
Height [Mean (Full Range); unit: meters] | 1.58 [1.55 to 1.63] | 1.65 [1.58 to 1.70] | 1.62 [1.55 to 1.70]
Weight [Mean (Full Range); unit: kgs] | 71.5 [62.8 to 76.4] | 76.1 [72.6 to 84.3] | 74.1 [62.8 to 84.3]
BMI [Mean (Full Range); unit: kg/m^2] | 28.6 [23.75 to 30.8] | 27.5 [25.06 to 29.83] | 28 [23.75 to 30.8]

OUTCOME MEASURES:

1. Primary Outcome: Post Surgical Drain Output in CCs
Description: Patient recorded, post operative drain output. Patients will track their 24-hour total drain output by recording the 24-hour total output at 10 am every day. If the output exceeds the drain capacity during the 24-hour interval but before the 10am empty time, the patient will empty the drain when full, record that output, allow the drain output to reaccumulate, and empty-record the drain output again at 10am or again when the output exceeds the drain capacity. The individual outputs recorded during the 24-hour interval will then be totaled to determine one output sum for the entire 24-hour time period between 10am time intervals. Each drain bulb will accommodate a maximum of 60cc of postoperative fluid. Drain removal will occur when output is less than 30 cc per drain in 24-hour period or eight weeks post-operatively.
Time Frame: Up to eight weeks post-operatively
Population: Data did not undergo analysis due to errors in data collection. Subjects were to have two 15 round Blake drains, however some of the subjects received French drains. Drain output was to be self recorded by the patient and was found to be inconsistent per data collection. The data was not analyzed due to small sample size and errors in the data collection process. As this study was a pilot, it was terminated for logistical concerns with these errors.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Participants With Post Operative Hematoma
Description: Patients will be monitored clinically at each post-operative visit for signs of post-operative hematoma or seroma. Each patient will be evaluated one week, three weeks, and eight weeks following their procedure to assess overall wound healing.
Time Frame: Up to 8 weeks postoperatively
Population: This is a count of the number of patients that experienced post operative hematoma.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 4 | 5
Participants | 0 | 1

3. Secondary Outcome: Number of Participants That Returned to the Operating Room
Description: Return to the operating room for evacuation post surgical operative hematoma or seroma assessed by clinical evaluation to include palpation for ballotable fluid collection and assessment of skin for a shiny/tight appearance suggestive of an underlying fluid collection.
Time Frame: Up to 8 weeks postoperatively
Population: This measure describes the number of patients in counts, that returned to the operating room for fluid collection.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

4. Secondary Outcome: Number of Days Until Drain Removal
Description: The number of days that the post surgical drains remain in place after the surgery. When less than 30 cc per drain in a 24-hour period, the participants are to call and schedule drain removal.
Time Frame: Up to 56 days post operatively.
Population: The average number of days that the participants endured the drains after surgery.
Measure: Mean (Full Range); unit: Days
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 4 | 5
Days | 16 [11 to 24] | 22 [15 to 39]

ADVERSE EVENTS:
Time Frame: 8 weeks postoperatively
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 4/4 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=4) | Group 2 (N=5)
Drain size (Surgical and medical procedures) | 4 (4) | 1 (5) — Error in drain size; 19" instead of required 15".
Error in number of sponges (Surgical and medical procedures) | 4 (4) | 2 (2) — Used less than 3 required sponges that were used to administer the interventional product vs saline.
Drain output (Surgical and medical procedures) | 3 (3) | 1 (1) — Error in documentation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT04902950/Prot_SAP_000.pdf